CLINICAL TRIAL: NCT03203902
Title: Comparative Effectiveness of Stress Management Using Psychoeducation Versus Therapeutic Touch for Formerly Homeless Adults With Mental Illness and Substance Use Histories
Brief Title: Comparative Effectiveness of Stress Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Sharon Gutman, Professor of Rehabilitation and Regenerative Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAR4338
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Stress
Keywords: Therapeutic touch; Post-traumatic Stress Disorder; Homeless
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Three arm, randomized controlled design
Who Masked: Participant
Masking Description: Participants receiving sham and authentic therapeutic touch will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psychoeducation and Therapeutic Touch (Active Comparator): 6-week psychoeducation group. The following 1-hour modules will be delivered:
  Week 1: Anger Management and Conflict Negotiation Week 2: Meditation and Breathing Techniques Week 3: Nutrition Week 4: Exercise, Leisure, and Recreation Week 5: Sleep Week 6: Wellness Recovery Action Plan (WRAP)
  Directly after the psychoeducation group is completed, 30-minute therapeutic touch will be administered.
  Interventions: Other: Psychoeducation and Therapeutic Touch
- Psychoeducation and Sham Therapeutic Touch (Placebo Comparator): 6-week psychoeducation group. The following 1-hour modules will be delivered:
  Week 1: Anger Management and Conflict Negotiation Week 2: Meditation and Breathing Techniques Week 3: Nutrition Week 4: Exercise, Leisure, and Recreation Week 5: Sleep Week 6: Wellness Recovery Action Plan (WRAP)
  Directly after the psychoeducation group is completed, 30-minute sham therapeutic touch will be administered.
  Interventions: Other: Psychoeducation and Therapeutic Touch
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Psychoeducation and Therapeutic Touch — 6-week, 1-hour psychoeducation group followed by 30-minute therapeutic touch
  Arms: Psychoeducation and Sham Therapeutic Touch; Psychoeducation and Therapeutic Touch

SUMMARY:
Many formerly homeless adults with chronic mental illness experience treatment resistant symptoms for which pharmaceutical agents and cognitive behavioral therapy are not effective. Although formerly homeless adults with chronic mental illness typically receive medical and psychiatric services to manage their illness, chronic stress and post-traumatic stress disorder (PTSD) acquired from homelessness are difficult to resolve and many adults experience relapse that can result in housing loss. Therapeutic touch is a complementary and alternative treatment that has been shown to be effective at reducing stress, anxiety, and pain in a variety of diagnoses including cancer, cardiac disease, chronic pain syndromes, and PTSD in veterans. In this study the investigators aim to determine whether a 30-minute therapeutic touch session combined with a conventional 1-hour psychoeducation group delivered over 6 weeks can more effectively reduce stress compared to conventional psychoeducation alone. The ability to reduce stress levels and maintain emotional equilibrium is critical for this population to manage illness symptoms effectively and stave off the incidence of relapse, rehospitalizations, and housing loss.

DETAILED DESCRIPTION:
In 2015, approximately 600,000 people were reported to be homeless on any given night in the United States and 1.6 million used homeless shelter services. One-third of homeless adults who received shelter services were diagnosed with chronic mental illness (e.g., schizophrenia, bipolar disorder, major depression) and two-thirds had substance use disorders.

Once housed in supportive living residences, formerly homeless adults with mental illness commonly continue to experience high levels of stress, anxiety, depression, and post-traumatic stress disorder (PTSD), despite receiving medical and psychiatric services. Stress that is not sufficiently addressed can frequently lead to rehospitalizations and subsequent loss of housing. Although stress has been successfully treated with anti-anxiety pharmaceuticals, cognitive behavioral therapies, and support groups in adults in the larger population, formerly homeless adults with chronic mental illness tend to experience greater treatment resistance to such interventions or respond positively for short intervals and then relapse.

One nonpharmacological intervention that has gained increasing support in the last two decades is therapeutic touch. Therapeutic touch, also referred to as healing touch and touch therapy, is a complementary and alternative treatment in which practitioners seek to alleviate or reduce pain, stress, or anxiety through direct hand contact with a client's bio- or energy field. A bio- or energy field is defined in quantum physics as an interconnected web of energy that surrounds living organisms and may regulate emotional states and physical health. Although the existence of energy fields is increasingly accepted in the scientific community, the precise roles of and mechanisms through which energy fields work are not understood. While eastern health practitioners have for centuries used therapies addressing energy fields-for example, acupuncture, acupressure, Ayurveda, qi gong-western practitioners have only begun using such therapies in the last century. The most common western names for energy field therapy are therapeutic touch, healing touch, Reiki, and touch therapy-all of which have growing bodies of evidence supporting their effectiveness in the reduction of stress, anxiety, and pain in various diagnostic populations including cancer, cardiovascular disease, and chronic pain syndromes.

Although there is evidence that therapeutic touch can help reduce symptoms of PTSD in veterans, and stress and anxiety in cancer and cardiac patients, little information exists about whether therapeutic touch can reduce stress in formerly homeless adults with chronic mental illness. The ability to reduce stress in formerly homeless adults may help them manage illness symptoms better and prevent relapse for longer intervals.

In this comparative effectiveness study, the investigators will provide a conventional stress management psychoeducation group to 20 participants. Ten of these 20 participants will additionally receive 30 minutes of therapeutic touch delivered in a group setting. The remaining 10 participants will receive 30 minutes of sham therapeutic touch delivered in a group setting. Ten additional participants will be allocated to a control group with no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Current supportive housing resident
* History of homelessness
* History of mental illness

Exclusion Criteria:

* Severe behavioral or anger management disorder

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Difference in Score on Perceived Stress Scale between pre- and post-intervention | baseline and 7 weeks
  5-point, 10-item Likert scale that takes approximately 5 minutes to complete

SECONDARY OUTCOMES:
Difference in Score on World Health Quality of Life Scale between pre- and post-intervention | baseline and 7 weeks
  5-point, 26-item scale that takes approximately 15 minutes to complete

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Gutman, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] US Department of Housing and Urban Development. (2015) 2015 Annual Homeless Assessment Report (AHAR) to Congress (November 2015). Retrieved from https://www.hudexchange.info/resources/documents/2015-AHAR-Part-1.pdf
- [Background] Treatment Advocacy Center. (2014) Eliminating barriers to the treatment of mental illness. How many individuals with a serious mental illness are homeless? Retrieved from http://www.treatmentadvocacycenter.org/problem/consequences-ofnon-treatment/2058
- [Background] Office of National Drug Control Policy. (n.d.) Chapter 3. Integrate treatment for substance use disorders into mainstream health care and expand support for recovery. Retrieved from https://www.whitehouse.gov/ondcp/chapter-integrate-treatment-forsubstance-use-disorders
- [Background] Lippert AM & Lee BA. Stress, coping, and mental health differences among homeless people. Sociological Inquiry. 2015 85(3), 343-374. doi:10.1111/soin.12080
- [Background] Lee CM, Mangurian C, Tieu L, Ponath C, Guzman D, Kushel M. Childhood Adversities Associated with Poor Adult Mental Health Outcomes in Older Homeless Adults: Results From the HOPE HOME Study. Am J Geriatr Psychiatry. 2017 Feb;25(2):107-117. doi: 10.1016/j.jagp.2016.07.019. Epub 2016 Aug 17. PMID 27544890
- [Background] Harvey PD, Rosenthal JB. Treatment resistant schizophrenia: Course of brain structure and function. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Oct 3;70:111-6. doi: 10.1016/j.pnpbp.2016.02.008. Epub 2016 Feb 27. PMID 26925705
- [Background] Roe CA, Sonnex C, Roxburgh EC. Two meta-analyses of noncontact healing studies. Explore (NY). 2015 Jan-Feb;11(1):11-23. doi: 10.1016/j.explore.2014.10.001. Epub 2014 Oct 23. PMID 25457442
- [Background] Meissner K, Koch A. Sympathetic Arousal during a Touch-Based Healing Ritual Predicts Increased Well-Being. Evid Based Complement Alternat Med. 2015;2015:641704. doi: 10.1155/2015/641704. Epub 2015 Jul 5. PMID 26236381
- [Background] Nourbakhsh MR, Bell TJ, Martin JB, Arab AM. The Effects of Oscillatory Biofield Therapy on Pain and Functional Limitations Associated with Carpal Tunnel Syndrome: Randomized, Placebo-Controlled, Double-Blind Study. J Altern Complement Med. 2016 Nov;22(11):911-920. doi: 10.1089/acm.2016.0083. Epub 2016 Aug 3. PMID 27487406
- [Background] Prakash S, Chowdhury AR, & Gupta, A. (2015). Monitoring the human health by measuring the biofield
- [Background] Anderson JG, Taylor AG. Effects of healing touch in clinical practice: a systematic review of randomized clinical trials. J Holist Nurs. 2011 Sep;29(3):221-8. doi: 10.1177/0898010110393353. Epub 2011 Jan 12. PMID 21228402
- [Background] Hammerschlag R, Marx BL, Aickin M. Nontouch biofield therapy: a systematic review of human randomized controlled trials reporting use of only nonphysical contact treatment. J Altern Complement Med. 2014 Dec;20(12):881-92. doi: 10.1089/acm.2014.0017. PMID 25181286
- [Background] Jain S, McMahon GF, Hasen P, Kozub MP, Porter V, King R, Guarneri EM. Healing Touch with Guided Imagery for PTSD in returning active duty military: a randomized controlled trial. Mil Med. 2012 Sep;177(9):1015-21. doi: 10.7205/milmed-d-11-00290. PMID 23025129
- [Background] Krucoff MW, Crater SW, Green CL, Maas AC, Seskevich JE, Lane JD, Loeffler KA, Morris K, Bashore TM, Koenig HG. Integrative noetic therapies as adjuncts to percutaneous intervention during unstable coronary syndromes: Monitoring and Actualization of Noetic Training (MANTRA) feasibility pilot. Am Heart J. 2001 Nov;142(5):760-9. doi: 10.1067/mhj.2001.119138. PMID 11685160
- [Background] Tabatabaee A, Tafreshi MZ, Rassouli M, Aledavood SA, AlaviMajd H, Farahmand SK. Effect of Therapeutic Touch in Patients with Cancer: a Literature Review. Med Arch. 2016 Apr;70(2):142-7. doi: 10.5455/medarh.2016.70.142-147. Epub 2016 Apr 1. PMID 27194823